CLINICAL TRIAL: NCT04394195
Title: sFlt1: a Biomarker of Organ Dysfunction in Critically-ill Patients With COVID-19?
Acronym: COVIDsFlt1
Status: Completed | Type: Observational
Sponsor: CHU de Reims (Other)
Responsible Party: Sponsor
Other Study IDs: PO20043*
Record Dates: First submitted 2020-05-16; First posted 2020-05-19 (Actual); Last update posted 2021-04-01 (Actual); Status verified 2021-03

CONDITIONS: CORONAVIRUS INFECTIONS
MeSH Terms: conditions — Coronavirus Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: None Retained — blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- patients with COVID-19 infection: patients with COVID-19 infection
  Interventions: Other: measurement of circulating sFlt1 concentration

INTERVENTIONS:
Other: measurement of circulating sFlt1 concentration — blood circulating sFlt1 concentration will be determined

SUMMARY:
Short description of the protocol intended for the lay public. Include a brief statement of the study hypothesis (Limit : 5000 characters) The management of critically-ill patients with organ failure due to COVID-19 represents a major healthcare burden. While endothelial inflammation has been reported in these patients, the pathophysiological mechanisms remain incompletely elucidated.

DETAILED DESCRIPTION:
Extended description of the protocol, including more technical information (as compared to the Brief Summary) if desired. Do not include the entire protocol; do not duplicate information recorded in other data elements, such as eligibility criteria or outcome measures. (Limit : 32 000 characters)

The soluble fms-like tyrosine kinase 1 (SFlt1) is the soluble form of VEGF-A receptor 1 (VEGFR1). By linking VEGF-A with a high affinity, sFlt1 blocks the VEGF-A / VEFR1 axis and impairs endothelial homeostasis. Its production increases during inflammation. We hypothesize that sFlt1 is upregulated and correlates with endothelial dysfunction and outcomes in critically-ill patients with COVID-19.

ELIGIBILITY:
Inclusion Criteria:

* Patient with documented COVID-19 (positive PCR)
* Hospitalized in University Hospital of Reims
* Patient or family who have previously consented

Exclusion Criteria:

* Patient <18 yo
* Patient not insured under the French social security

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All adult patients with COVID-19 hospitalized in University Hospital of Reims
Sampling Method: Non-Probability Sample
Enrollment: 72 (Actual)
Dates: Start 2020-04-03 (Actual); Primary Completion 2020-05-01 (Actual); Study Completion 2020-09-01 (Actual)

PRIMARY OUTCOMES:
Association between concentration of circulating sFlt1 and use of vasopressor | 14 days

CONTACTS AND LOCATIONS:
Locations (1):
- Chu Reims, Reims, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Dupont V, Kanagaratnam L, Goury A, Poitevin G, Bard M, Julien G, Bonnivard M, Champenois V, Noel V, Mourvillier B, Nguyen P. Excess Soluble fms-like Tyrosine Kinase 1 Correlates With Endothelial Dysfunction and Organ Failure in Critically Ill Coronavirus Disease 2019 Patients. Clin Infect Dis. 2021 May 18;72(10):1834-1837. doi: 10.1093/cid/ciaa1007. PMID 32672790